CLINICAL TRIAL: NCT01127152
Title: Assessment of Automatic Relays by Intensive Basis Advantage Compared With Manual Relays, on the Hypotension Risks, During Noradrenalin Administration
Acronym: ARIBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD 010-09
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hypotension
Keywords: Noradrenalin relays; Automatic relays; Manual relays; Hypotension; Intensive care unit
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automatic relays (Active Comparator): Automatic relays of noradrenalin using intensive basis.
  Interventions: Procedure: Measure of arterial pressure
- Manual relays (Active Comparator): Relays of noradrenalin using manual method
  Interventions: Procedure: Measure of arterial pressure

INTERVENTIONS:
Procedure: Measure of arterial pressure — Measure of arterial pressure will occur every five minutes during the thirty minutes before the relay and during the fifteen minutes after the relay.

SUMMARY:
Circulatory failures are the main cause of admissions in the intensive care unit. It is recommended to prescribe to these patients an intravenous injection of catecholamine to correct this dysfunction and to keep an hemodynamic stability. Electric pumps are used to administrate a continuous flow of drugs to patient. When a syringe of drugs ends, it is replaced by a full syringe, it is named "relay". This change may cause a flow interruption and hypotension.

In the intensive care unit at departmental hospital (CHD) Vendee, the manual relays used in common practice will cause hemodynamic instabilities : hypotensions in 20% cases. Since 4 years, new devices are also used to make the relays. It is "smart pumps" allowing to manage automated the drug delays. This new method allows to not interrupt the drug flow. It could reduce the occurence of hypotension. A 50% decrease of relative number of hypotension will show that the use of automatic method is the most sure medical strategy.

Our study want to compare manual and automatic method watching the variations of medium arterial pressure (MAP) during the fifteen minutes after the relay compared to baseline (MAP before the relay). Noradrenalin is the catecholamine most administrated so we choose to study only the relay for this drug.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years,
* Patient receiving only noradrenalin as catecholamine,
* Collection of patient's non-objection or his trustworthy person, if appropriate.

Exclusion Criteria:

* Pregnant or breast feeding patient,
* Patient receiving an other treatment on the catecholamine way,
* No affiliation at a social security,
* Refusal of patient's trustworthy person or parent, if the patient is unable to give his non-objection.
* Refusal of patient's participation when he is conscious,
* Subjects deprived of liberty, under guardianship, hospitalized in a health facility or social or hospitalized without their consent,
* Patients with secreting tumor, kind pheochromocytoma ou carcinoid tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Hypotension occurence defined as a decrease of 20% of the medium arterial pressure(MAP) between the baseline (MAP before the relay) and the minimal MAP in the fifteen minutes after the relay. | every five minutes during the thirty minutes before the relay, during the fifteen minutes after the relay

SECONDARY OUTCOMES:
Number of relays where the medium arterial pressure (MAP) is decreased by 10% compared to baseline | every five minutes during the thirty minutes before the relay, during the fifteen minutes after the relay
Number of relays where the medium arterial pressure (MAP) is inferior to 50 millimeter of mercury (mmHg) | during the fifteen minutes after the relay
Number of hypotension in patients whose dose of noradrenalin is > 0,5 gamma/kg/min | every five minutes during the thirty minutes before the relay, during the fifteen minutes after the relay

CONTACTS AND LOCATIONS:
Overall Officials: Jean Reignier, MD, Principal Investigator — CHD Vendée
Locations (1):
- CHD Vendée, La Roche-sur-Yon, Vendée, France

REFERENCES:
- [Result] Greau E, Lascarrou JB, Le Thuaut A, Maquigneau N, Alcourt Y, Coutolleau A, Rousseau C, Erragne V, Reignier J. Automatic versus manual changeovers of norepinephrine infusion pumps in critically ill adults: a prospective controlled study. Ann Intensive Care. 2015 Dec;5(1):40. doi: 10.1186/s13613-015-0083-7. Epub 2015 Nov 14. PMID 26577132